CLINICAL TRIAL: NCT03142204
Title: Study of the Kinetics, Dosimetry and Safety of [18F]F-AraG (VisAcT), a Positron Emission Tomography Tracer for Imaging the Activation of the Immune System in Cancer Patients Who Have Received or Are Expected to Receive Immunotherapy and/or Radiation Therapy
Brief Title: [18F]FAraG PET Imaging for Analysis of Biodistribution in Cancer Patients Expected to Undergo Immunotherapy and/or Radiation Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CellSight Technologies, Inc. (Industry)
Collaborators: UCSF Imaging Center at China Basin (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-14488
Record Dates: First submitted 2017-05-01; First posted 2017-05-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: [18F]F-AraG — Single dose IV injection of [18F]F-AraG for each imaging day.

SUMMARY:
This is a Phase 1 study is to visualize biodistribution of a PET tracer called [18F]F-AraG (VisAcT) in cancer patients expected to undergo immunotherapy and/or radiation therapy.

DETAILED DESCRIPTION:
This is an exploratory Phase 1, prospective study assessing the biodistribution and radiation dosimetry of the Positron Emission Tomography [18F]FAraG (VisAcT) in cancer patients selected for immunotherapy and/or radiation therapy. Each patient may have up to two [ 18F]FAraG PET imaging sessions, a baseline scan and a post start of immunotherapy scan. For each imaging session, patients will receive a single injection of [18F]FAraG and undergo a whole-body PET scans an hour after injection of the tracer. Following each imaging session, the patient will be called within 72 hours to note any side effects.

Optional - Blood samples may be collected at up to 9 time points post-injection to analyze whole-blood/plasma time activity of [18F]FAraG in addition an urine sample may be collected post scan.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients with identified tumor mass
* Cancer patients expected to undergo immunotherapy and/or radiation therapy

Exclusion Criteria:

* Under the age of 18
* Pregnant women
* Women who are breastfeeding
* Individuals with known or suspected substance abuse
* Individuals unable or unwilling to comply with the study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Visualize biodistribution of the PET tracer [18F]F-AraG pre-immunotherapy | Up to 6 weeks before immunotherapy is administered
  Whole-body [18F]F-AraG PET scan will be performed after intravenous injection of the PET tracer.consecutive time points the day of the intravenous injection of the PET tracer.
Visualize biodistribution of the PET tracer [18F]F-AraG post start of immunotherapy | Up to 12 weeks after start of immunotherapy
  Whole-body [18F]F-AraG PET scan will be performed after intravenous injection of the PET tracer.

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Flavell, M.D., Ph.D., Principal Investigator — UCSF Department of Radiology & Biomedical Imaging
Locations (1):
- UCSF Imaging Center at China Basin, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No